CLINICAL TRIAL: NCT00371176
Title: A Placebo-Controlled Trial of D-Cycloserine and Exposure Therapy for Combat-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORD-NIMH-20061
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2013-12

CONDITIONS: Combat Disorders; Stress Disorders, Post-Traumatic
Keywords: Cognitive Behavior Therapy; Cognitive enhancers; Combat Disorders; D-Cycloserine; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Implosive Therapy; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-Cycloserine (Experimental): Brief imaginal exposure therapy plus DCS pill
  Interventions: Behavioral: Exposure therapy; Drug: D-Cycloserine
- Placebo (Placebo Comparator): Brief imaginal exposure therapy plus Placebo pill
  Interventions: Behavioral: Exposure therapy; Other: Placebo pill

INTERVENTIONS:
Behavioral: Exposure therapy — A manualized form of treatment that involves vividly visualizing indexed trauma with the guidance of a therapist
Drug: D-Cycloserine — A partial NMDA agonist that has been shown in human trials to facilitate and strengthen extinction with CBT.
  Arms: D-Cycloserine
Other: Placebo pill
  Arms: Placebo

SUMMARY:
The primary aim of this project is to examine whether administration of D-Cycloserine (DCS), a partial N-methyl-D-aspartate (NMDA) receptor agonist that has been shown to facilitate fear extinction, enhances the therapeutic benefit of exposure-based cognitive behavioral therapy (CBT) in OEF/OIF veterans with PTSD.

DETAILED DESCRIPTION:
War-zone-related posttraumatic stress disorder (PTSD) is a major psychiatric disorder that includes specific disabling symptoms and impairments that interfere with a soldier's ability to do his or her job. There is strong evidence for cognitive behavior therapy (CBT) in treating PTSD in civilians, which suggests a prescription for returning veterans, but approximately 40% of patients retain a PTSD diagnosis (e.g., Foa et al., 1999) and drop-out rates are ~25%. It is imperative to develop novel evidence-based early interventions that are more acceptable to recent veterans and less draining of treatment resources. If CBT can be shortened and its efficacy boosted by cognitive enhancers then it is more likely that soldiers will get the most efficacious treatments for acute stress and PTSD. Our aim is to develop a program that is brief and effective, but will have long-term benefits for veterans by virtue of its greater amenability to self-management and treatment adherence beyond the therapy context.

This study is a randomized, controlled, double-blind treatment trial comparing CBT plus DCS to CBT plus placebo. Participants will be 68 OEF/OIF veterans with PTSD randomly assigned to CBT plus DCS or CBT plus placebo. Procedures to screen subjects prior to randomization include a detailed phone screen, administration and collection of questionnaires, a medical assessment, and two baseline structured clinical interviews. Following randomization, both groups will receive the identical 6 session exposure-based CBT protocol. The DCS-augmented group will receive 50 mg of DCS 30 minutes prior to the four CBT sessions involving imaginal exposure, whereas the placebo-augmented group will receive a placebo pill prior to these sessions. Assessment interviews conducted by independent evaluators will occur at pre-treatment, post-treatment, and at 3, and 6-month follow-up. Self-report measures will also be administered at screening, throughout the 6 weeks of treatment, and at 3- and 6- month follow up.

Comparison(s): OEF/OIF veterans with PTSD treated with CBT plus DCS, compared to OEF/OIF veterans with PTSD treated with CBT plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years of age or older who served in Operation Iraqi Freedom or Operation Enduring Freedom (OIF/OEF) and who have a primary diagnosis (designated by the patient as the most important source of distress of PTSD.
* Willingness and ability to comply with the requirements of the study protocol.

Exclusion Criteria:

A lifetime history of:

* bipolar disorder
* schizophrenia
* psychosis
* delusional disorders or obsessive-compulsive disorder
* organic brain syndrome
* cognitive dysfunction that could interfere with capacity to engage in therapy
* a history of substance or alcohol dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
* Patients with significant suicidal ideation or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate services.
* Patients must be off concurrent psychotropic medication (e.g., antidepressants, anxiolytics, beta blockers) for at least 2 weeks prior to initiation of randomized treatment.
* Serious medical illness or instability for which hospitalization may be likely within the next year.
* Patients with a current or past history of seizures
* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception (e.g., intra uterine device, oral contraceptives, barrier devices, condoms and foam, or implanted progesterone rods stabilized for at least 3 months).
* Any concurrent psychotherapy initiated within 3 months of baseline, or ongoing psychotherapy of any duration specifically targeting PTSD is excluded. General supportive therapy initiated > 3 months prior is acceptable.
* Patients with seizures or ongoing severe cognitive impairment that compromised mental status.
* Patients receiving Isoniazid.
* Patients unable to understand study procedures and participate in the informed consent process.
* Patients with a history of renal insufficiency (creatinine clearance less than 50 mL/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-10; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett T. Litz, PhD, Principal Investigator — VA Boston Health Care System
Locations (1):
- VA Boston Health Care System, Boston, Massachusetts, United States

REFERENCES:
- [Result] Litz BT, Salters-Pedneault K, Steenkamp MM, Hermos JA, Bryant RA, Otto MW, Hofmann SG. A randomized placebo-controlled trial of D-cycloserine and exposure therapy for posttraumatic stress disorder. J Psychiatr Res. 2012 Sep;46(9):1184-90. doi: 10.1016/j.jpsychires.2012.05.006. Epub 2012 Jun 12. PMID 22694905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was 2007 to 2011. Participants were recruited through VA clinician referrals and public advertising (e.g., flyers and radio ads).
Groups:
- D-Cycloserine Plus Exposure: Treatment entailed six 60-90 minute sessions. Session 1 focused on psychoeducation and building of rapport, sessions 2-5 of brief imaginal exposure therapy plus a 50 mg DCS pill 30 minutes prior to each session, and session 6 consisted of a review of treatment gains, discussion of relapse-prevention strategies, and termination.
- Placebo Plus Exposure: Treatment entailed six 60-90 minute sessions. Session 1 focused on psychoeducation and building of rapport, sessions 2-5 of brief imaginal exposure therapy plus a placebo pill 30 minutes prior to each session, and session 6 consisted of a review of treatment gains, discussion of relapse-prevention strategies, and termination.
Period: Overall Study
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Started | 13 | 13
Completed Treatment | 10 | 9
Completed | 8 | 5
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- D-Cycloserine Plus Exposure: Brief imaginal exposure therapy plus DCS pill
- Placebo Plus Exposure: Brief imaginal exposure therapy plus Placebo pill
- Total: Total of all reporting groups
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.77 (9.85) | 31.62 (9.10) | 32.19 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale-IV
Description: A 17-item, semi-structured interview of PTSD symptoms. The range of scores is 0-136, with a higher value representing a worse outcome.
Time Frame: Pre Intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 13 | 13
units on a scale | 69.85 (23.24) | 73.38 (16.35)

2. Secondary Outcome: PTSD Checklist
Description: A 17-item, self-report measure of PTSD symptoms. The range of scores is 17-85, with a higher value representing a worse outcome.
Time Frame: Pre Intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 13 | 13
units on a scale | 37.85 (8.76) | 39.00 (8.77)

3. Secondary Outcome: PTSD Checklist
Description: as for outcome 2
Time Frame: Post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 13 | 13
units on a scale | 34.11 (21.09) | 24.18 (14.95)

4. Primary Outcome: Clinician Administered PTSD Scale-IV
Description: as for outcome 1
Time Frame: Post Intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 13 | 13
units on a scale | 72.33 (28.68) | 53.73 (26.22)

5. Primary Outcome: Clinician Administered PTSD Scale-IV
Description: as for outcome 1
Time Frame: 3 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 9 | 11
units on a scale | 62.57 (32.17) | 58.20 (26.17)

6. Primary Outcome: Clinician Administered PTSD Scale-IV
Description: as for outcome 1
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 9 | 11
units on a scale | 62.20 (32.17) | 55.50 (27.02)

7. Secondary Outcome: PTSD Checklist
Description: as for outcome 2
Time Frame: 3 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 9 | 11
units on a scale | 33.29 (14.68) | 26.91 (16.40)

8. Secondary Outcome: PTSD Checklist
Description: as for outcome 2
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 9 | 11
units on a scale | 29.20 (13.16) | 27.25 (15.83)

9. Secondary Outcome: Beck Depression Inventory
Description: A 21-item, self-report measure of depression symptoms. The range of scores is 0-63, with a higher value representing a worse outcome.
Time Frame: Pre intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 13 | 13
units on a scale | 24.85 (15.31) | 21.48 (9.24)

10. Secondary Outcome: Beck Depression Inventory
Description: as for outcome 9
Time Frame: Post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 13 | 13
units on a scale | 28.56 (16.25) | 14.18 (10.81)

11. Secondary Outcome: Beck Depression Inventory
Description: as for outcome 9
Time Frame: 3 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 9 | 11
units on a scale | 24.57 (14.43) | 13.90 (10.59)

12. Secondary Outcome: Beck Depression Inventory
Description: as for outcome 9
Time Frame: 6 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Number analyzed (Participants) | 9 | 11
units on a scale | 22.25 (17.73) | 15.38 (11.43)

ADVERSE EVENTS:
Arm/Group | D-Cycloserine Plus Exposure | Placebo Plus Exposure
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
The study experienced sustained recruitment difficulties, ultimately recruiting a smaller number of participants (N=26) than originally projected (N=68).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No